## Statistical Analysis Plan

**Title** 

Temporary Aortic Occlusion with the Abdominal Tourniquet for Refractory Postpartum Haemorrhage: A Proof-of-Concept Study in a War-Affected Region

### Version

1.0

### **Date**

November 1, 2024

## **Principal Investigators**

Dr. Yevheniia Poliakova, MD, PhD — Olexandrivska Hospital, Zaporizhzhia

Dr. Viktor Oshovskyy, MD, PhD, DMSc — Uniklinika Medical Centre, Kyiv

### Institution

Olexandrivska Hospital, Zaporizhzhia, Ukraine

## **Ethics Approval**

Approved by Olexandrivska Hospital Ethics Committee (Approval number: 2024/EC/128094)

# 1. Objectives

## 1.1. Primary Objective

• To assess the feasibility and preliminary effectiveness of the AAJT-S device in controlling refractory postpartum haemorrhage (PPH) due to uterine atony in a waraffected, resource-limited setting.

## 1.2. Secondary Objectives

- To evaluate the safety profile of the AAJT-S device (device-related complications, thrombotic events, ischemic injuries, infection).
- To assess the duration of bleeding control and time to definitive surgical intervention.

# 2. Study Design

- **Design**: Prospective, single-center, open-label, non-randomized, proof-of-concept study.
- Sample Size: 4 patients
- **Analysis Type**: Descriptive statistics only. No inferential testing or hypothesis-driven comparisons will be performed due to small sample size and exploratory nature.

# 3. Analysis Populations

- Full Analysis Set (FAS): All patients who received AAJT-S for refractory PPH.
- **Safety Population**: Identical to FAS; all patients who underwent device placement and were monitored until discharge.

## 4. Variables

### 4.1. Baseline Characteristics

- Age (years)
- Gravida and Para
- Gestational Age at delivery (weeks + days)

### 4.2. Effectiveness Outcomes

- Time to bleeding control (minutes from inflation to cessation of visible bleeding)
- Total duration of AAJT-S placement (minutes)
- **Definitive surgical interventions performed** (Yes/No; type of procedure)
- Total cumulative measured blood loss (CMBL) (mL)
- Need for blood transfusion (Yes/No; units PRBC and FFP)

## 4.3. Safety Outcomes

- Thrombotic events (Yes/No)
- **Ischemic injury** (Yes/No)
- Device-related complications (e.g., skin necrosis, incorrect placement)
- Infectious complications (e.g., sepsis, wound infection)
- **Readmissions** or complications during postpartum follow-up (Yes/No)

# 5. Statistical Methods

### 5.1. Descriptive Analysis

- Continuous variables: summarized using median, range (min-max).
- Categorical variables: presented as counts and percentages.

## 5.2. No inferential statistics

- Given the small sample size, **no hypothesis testing**, **p-values**, or **confidence intervals** will be calculated.
- No missing data imputation will be applied. All available data will be included in descriptive summaries.

### **5.3. Software**

• All analyses will be performed using **Microsoft Excel (Version 16.83)**. No specialized statistical software was used due to the simplicity and exploratory nature of the data.

# 6. Data Handling and Quality Assurance

- Clinical data were extracted from patient medical records and entered manually into a study-specific Excel spreadsheet.
- Double-checking was conducted for critical variables (e.g., blood loss, time intervals) by both study investigators.

# 7. Limitations

- Small sample size prevents generalizability.
- No control group.
- Estimates of blood loss may be subject to observer bias.